CLINICAL TRIAL: NCT03742323
Title: Phase I-II Unmasked, Non-randomized Study Evaluating the Role of Idelalisib in Patients With Acute Lymphoblastic Leukemia (ALL) That is Relapsing or Refractory to Other Treatments, and in Older Patients With ALL for Whom Conventional Treatments Are Not Recommended
Brief Title: REALIB-LLA-2017: Idelalisib in Patients With Acute Lymphoblastic Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Because of low recruitment
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REALIB-LLA-2017
Record Dates: First submitted 2018-11-13; First posted 2018-11-15 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — idelalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Idelalisib (Experimental)
  Interventions: Drug: Idelalisib

INTERVENTIONS:
Drug: Idelalisib — Idelalisib Dose: 100, 150, 200 or 300 mg (in four cohorts of six patients each).
  Other Names: CAL-101

SUMMARY:
This study will attempt to confirm the hypothesis that Idelalisib may represent a new therapeutic alternative for patients with ALL in a set of particularly complex scenarios: relapsed, refractory to conventional treatments, and old age. For this reason, the primary objective is the overall response rate [ORR, defined as complete response (CR) or CR with partial hematologic recovery (CRh) and response duration (RD) in adult patients with relapsed or refractory ALL, or in adult ALL patients who are not suitable for treatment with conventional therapies.

DETAILED DESCRIPTION:
Phase I-II multi-site, exploratory, interventional, unmasked, non-randomized, single arm clinical trial. A single drug will be administered in four different, increasing doses to four consecutive cohorts.

The first phase of the study will focus on determining the most effective and tolerated dose of the study drug. The second phase will follow patients to the end to evaluate the safety of the drug.

The dose escalation will be decided by the Study Coordinator, who will evaluate and assess each cohort. Once the cohort of 6 patients is complete, the Coordinator will evaluate patients and, based on the tolerability and efficacy obtained, will decide whether to proceed with the dose escalation, or whether to end the trial The study will remain open until the overall number of participants is achieved; §progressive dose increases (PI) will be discontinued if dose-limiting toxicity (DLT) is observed in more than two patients in the previous cohort, *PI of the dose will only continue (for the third cohort) if at least two patients in the first two cohorts achieve the overall response rate (ORR), that is, complete response (CR) at four weeks from initiation of treatment; ** the study will only move on to the fourth cohort if CR is achieved in at least one of the six patients in the third cohort at four weeks from initiation of treatment; ***microscopy/cytofluorometry; ****complete blood count, microscopy, biochemistry; *****as long as there is no relapse, treatment will continue after the end of the study (planned for 24 months after the start of recruitment); AE, adverse events

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* B-cell precursor ALL, in any of the following cases:

  * Second or subsequent relapses [including after hematopoeitic stem cell transplantation (HSCT)] in patients who are ineligible for subsequent HSCT.
  * Resistance to at least two lines of treatment. Line of treatment is understood as initial treatment y salvage therapy after the first relapse (that may include HSCT).
  * Older adult patients (aged >65 years) for whom standard therapies are not clinically advisable.
* In patients with Ph+ ALL, failure after receiving at least two treatments with different TKIs (tyrosine kinase inhibitors): imatinib, dasatinib or ponatinib, in patients who are ineligible for subsequent HSCT.
* ECOG between 0 and 2.
* Aspartate transaminase (AST) and alanine aminotransferase (ALT) values < two times the upper limit of normal (ULN) and total bilirubin 2 mg/dL.
* Creatinine <2 mg/dL
* More than 10% blasts in bone marrow in the two weeks prior to the start of the trial.
* Women of childbearing potential: must agree to practice abstinence (abstain from having heterosexual sexual relations/contact) or to use one highly effective birth control method (failure rate less than 1%) during the treatment period and for at least 28 day after the last dose of Idelalisib .
* A woman is considered able to conceive if she is menstruating, is not post-menopausal (≥12 consecutive months without menstruation for no cause other than menopause) and who has not undergone surgical sterilization (removal of ovaries or uterus).
* Examples of birth control methods with a <1% yearly failure rate include bilateral tubal ligation, vasectomy, proper use of hormonal contraceptives that prevent ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
* The feasibility of sexual abstinence should be evaluated with respect to the duration of the trial and the patient's normal lifestyle preferences. Periodic abstinence (for example, the calendar method, ovulation, symptothermal or post-ovulation methods) and the withdrawal method are not acceptable birth control methods.
* Male patients: must agree to practice abstinence (abstain from heterosexual sexual relations) or use birth control methods, and agree to not donate sperm, as defined below:
* With female partners of childbearing capacity or pregnant female partner, men must practice total abstinence or use a condom plus one additional birth control method which, combined, have a failure rate of <1% per year during the treatment period, and for at least 4 months after the last dose of Idelalisib to avoid exposure to the fetus. Men must not donate sperm during this same time period.
* The feasibility of sexual abstinence should be evaluated with respect to the duration of the trial and the patient's lifestyle preferences. Periodic abstinence and the withdrawal method are not acceptable birth control methods.

Exclusion Criteria:

* Isolated central nervous system relapse.
* Patients planning to undergo HSCT.
* Any active systemic fungal, bacterial, or viral infection at the time of inclusion in the study.
* Grade II-IV active diarrhea.
* Grade II-IV active liver toxicity.
* Previous treatment with other PI3K/mTOR inhibitors.
* Taking any other experimental drug at the time of entering the trial. Patients who have completed a 4-week washout period will be permitted to enrol in the trial.
* Taking any antineoplastic drugs at the time of entering the trial (an exception is made for patients being treated with hydroxyurea or glucocorticoids. Use of these drugs is allowed up to 24 hours before initiating treatment with Idelalisib ).
* Patients being treated with moderate or potent CYP3A4 inhibitors or inducers.
* Patients with Stevens-Johnson Syndrome and toxic epidermal necrolysis.
* Patients with active chronic hepatitis, including viral hepatitis.
* Patients with HIV.
* Medical history of pneumonitis or any baseline lung disorder that, in the investigator's opinion, might worsen the patient's prognosis in the event of opportunistic pneumonia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2020-06-02 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | 6 months
  overall response rate (ORR), defined as CR (blasts in bone marrow aspiration <5%; neutrophils >1x109/L and platelets>100x109/L in peripheral blood) or CR with partial hematologic recovery (RCh) (blasts in bone marrow aspiration <5%; neutrophils<1x109/L and/or platelets <100x109/L in peripheral blood).
Response duration | 6 months
  Time to response duration

SECONDARY OUTCOMES:
Overall Response Rate in subgroups | 6 months
  Determine ORR in distinct subgroups of ALL (Ph+ and Ph-).
Determine progression free survival (PFS). | 6 months
  Time to progression
Determine overall survival (OS). | 24 months
  Time of overall survival
Percentage of Adverse Events | 6 months
  Safety

CONTACTS AND LOCATIONS:
Locations (12):
- Spain (12):
  - Hospital ICO Badalona, Badalona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Vall d'Hebrón, Barcelona
  - Hospital ICO Hospitalet, L'Hospitalet de Llobregat
  - Hospital 12 de Octubre, Madrid
  - H. Virgen de la Victoria, Málaga
  - H. Morales Meseguer, Murcia
  - Hospital Clinico de Salamanca, Salamanca
  - Hospital Marques de Valdecilla, Santander
  - H. Universitario Virgen de Rocío, Seville
  - Hospital Clínico Valencia, Valencia
  - Hospital Universitario y Politécnico la Fe, Valencia

IPD SHARING:
Plan to Share IPD: Undecided